CLINICAL TRIAL: NCT05253326
Title: The Effect of Progressive Muscle Relaxation Exercises on Pain and Disability After Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Eda Polat, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulMU10
Record Dates: First submitted 2022-02-08; First posted 2022-02-23 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Lumbar Surgery; Progressive muscle relaxation; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercises Group (Experimental): Patients will be taught Progressive Muscle Relaxation Exercises before the surgery and will be applied twice a week for 2 months after the surgery.
  Interventions: Other: Progressive Muscle Relaxation Exercises
- Control Group (No Intervention): Patients in the control group will receive standard care that includes all medical and non-medical treatments in the hospital.

INTERVENTIONS:
Other: Progressive Muscle Relaxation Exercises — It is among the relaxation techniques that require the active participation of the individual.
  Arms: Exercises Group

SUMMARY:
This study was planned as a randomized controlled experimental study to determine the effect of progressive muscle relaxation exercises on pain and disability in patients undergoing spinal surgery.

DETAILED DESCRIPTION:
Low back pain is not a disease in itself, but a symptom with many causes. The term "low back pain" means pain felt close to the midline of the lumbar or sacral region. It is a common problem in the society that causes loss of workforce and is accepted as a common cause of disability (functional limitation). Vertebral compression fractures, degenerative joint disease, spinal stenosis and various mechanical disorders are among the causes of low back pain. Although due to other pathologies, the general opinion is that lumbar disc prolapses often suppress or irritate one or more nerve roots in the lumbosacral region, causing pain that radiates to certain areas of the hips or legs. This pain is defined as lumbosacral radiculopathy. Although lumbosacral radiculopathy is treated conservatively in many patients, surgery is a common option in patients with persistent symptoms. The aim of surgical treatment methods such as discectomy, laminectomy, foraminotomy and spinal fusion is to release the neural structures by removing the herniated disc that compresses the nerve root and dura. Although there are various outcomes to measure the success of treatment after lumbar disc surgery, reduction of pain and returning to normal activities remain the main goals for patients. In the studies performed, it was determined that almost every patient had low back and leg pain, low quality of life scores and high disability scores before the surgery, while it was determined that there was an improvement in pain and other areas after the surgery. However, in the literature, complete relief after surgery is rarely seen, and symptoms persist in patients; It is stated that the severity varies from minor and non-irritating to severe and debilitating. Persistent and recurrent radicular pain after lumbar surgery is often associated with compression of the nerve roots. Zanoli et al. (2001) found that after surgical interventions for degenerative lumbar spine diseases, tolerable pain continued in the same way or increased in the 4th and 12th months postoperatively. Häkkinen et al. (2004) found that although there was improvement in postoperative back and leg pain, 25% of the patients still had moderate or severe leg pain at the 2nd month postoperatively, and approximately 30% perceived moderate or severe disability. Similarly, Lee et al. (2017) also found that although there was an improvement in the level of pain after surgery, the pain continued at a moderate level in the 3rd, 6th and 12th months. Continuing pain, motor deficits and decreased functional capacity after lumbar disc surgery may also cause loss of work force. In a study on the subject, it was determined that 80% of the patients re-reported due to pain or retired early after a 2-month routine health report after lumbar disc surgery. Controlling pain is important in terms of relaxation of the individual, increasing the quality of life, reducing complications and shortening the length of hospital stay. Pharmacological and non-pharmacological methods are used in the control of pain. One of the non-pharmacological methods is "relaxation". Passive relaxation, biofeedback, autogenic relaxation, basic breathing exercises, and progressive relaxation exercises (PRE) are among the relaxation techniques that require the active participation of the individual. Relaxation therapy has recently become an integral part of the care of individuals with chronic diseases due to its benefits such as reducing anxiety and stress, distracting attention from pain, relieving muscle tension and contractions, facilitating sleep, reducing fatigue and sensitivity to pain. With relaxation therapy, individuals can notice the tensions in their bodies, control their muscles, and learn to relax and relax tense parts of the body. One of the simplest and easiest to learn relaxation techniques is progressive relaxation exercises. These exercises are a series of procedures involving deep breathing and stretching and relaxation cycles in 50 different muscle groups to increase awareness of muscle tension in the body and learn to release these muscles. The technique promotes the systematic relaxation of the main muscle groups of the body for the purpose of physical and mental relaxation, reduction of response to stress, reduction of skeletal muscle contractions and the sensation of pain. In the literature, there are many studies related to progressive relaxation exercises and pain in different patient groups. In studies on musculoskeletal pain, it has been shown that progressive relaxation exercises significantly reduce the pain of patients with chronic neck pain (Lauche et al. 2013), and have a significant effect on pain, stress and disability levels in patients with chronic low back pain. In a systematic review study, it is stated that PRE is effective in reducing chronic low back pain and improving functional status. No study has been found examining the effect of PRE on postoperative pain and disability in patients undergoing lumbar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone spinal surgery (such as Discectomy, Laminectomy, Spinal fusion, Foraminatomy),
* 18 years of age or older
* Agreeing to apply progressive relaxation exercises and willing and willing to participate in the study,
* Having no medically diagnosed health problems (neurological, psychiatric, orthopedic) that will prevent learning and practicing progressive muscle relaxation exercises,
* Patients who do not know and practice progressive relaxation exercises before will be included in the study.

Exclusion Criteria:

* Patients who will undergo emergency surgery,
* Do not want to apply progressive relaxation exercises,
* Do not apply them as desired during the working process,
* Those have health problems (neurological, psychiatric, orthopedic) that may affect their ability to do the exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Progressive Muscle Relaxation Exercises | 12 months
  Visual Analogue Scale scores will decrease after progressive muscle relaxation exercises. The highest score that can be obtained from the visual analog scale is 10 and the lowest 0. As the higher score is obtained, the patient's pain will increase, and the result is evaluated as bad.
Progressive Muscle Relaxation Exercises | 12 months
  Roland-Morris Disability Questionnaire will decrease after progressive muscle relaxation exercises.There will be a total score between 0-24. A high score indicates severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan 2. Abdülhamid Han Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be shared with other researchers by holding a meeting after the data collection is completed.

REFERENCES:
- [Background] Akmese ZB, Oran NT. Effects of Progressive Muscle Relaxation Exercises Accompanied by Music on Low Back Pain and Quality of Life During Pregnancy. J Midwifery Womens Health. 2014 Sep-Oct;59(5):503-9. doi: 10.1111/jmwh.12176. Epub 2014 Jun 25. PMID 24965313
- [Background] Atya AM. The validity of spinal mobility for prediction of functional disability in male patients with low back pain. J Adv Res. 2013 Jan;4(1):43-9. doi: 10.1016/j.jare.2012.01.002. Epub 2012 Feb 16. PMID 25685400
- [Background] Casser HR, Seddigh S, Rauschmann M. Acute Lumbar Back Pain. Dtsch Arztebl Int. 2016 Apr 1;113(13):223-34. doi: 10.3238/arztebl.2016.0223. PMID 27120496
- [Background] Chen YL, Francis AJ. Relaxation and imagery for chronic, nonmalignant pain: effects on pain symptoms, quality of life, and mental health. Pain Manag Nurs. 2010 Sep;11(3):159-68. doi: 10.1016/j.pmn.2009.05.005. Epub 2009 Sep 8. PMID 20728065
- [Background] Fekete TF, Haschtmann D, Kleinstuck FS, Porchet F, Jeszenszky D, Mannion AF. What level of pain are patients happy to live with after surgery for lumbar degenerative disorders? Spine J. 2016 Apr;16(4 Suppl):S12-8. doi: 10.1016/j.spinee.2016.01.180. Epub 2016 Feb 2. PMID 26850172
- [Background] Hasenbring MI, Plaas H, Fischbein B, Willburger R. The relationship between activity and pain in patients 6 months after lumbar disc surgery: do pain-related coping modes act as moderator variables? Eur J Pain. 2006 Nov;10(8):701-9. doi: 10.1016/j.ejpain.2005.11.004. Epub 2006 Jan 19. PMID 16426878
- [Background] Kucukdeveci AA, Tennant A, Elhan AH, Niyazoglu H. Validation of the Turkish version of the Roland-Morris Disability Questionnaire for use in low back pain. Spine (Phila Pa 1976). 2001 Dec 15;26(24):2738-43. doi: 10.1097/00007632-200112150-00024. PMID 11740366
- [Background] Lauche R, Materdey S, Cramer H, Haller H, Stange R, Dobos G, Rampp T. Effectiveness of home-based cupping massage compared to progressive muscle relaxation in patients with chronic neck pain--a randomized controlled trial. PLoS One. 2013 Jun 7;8(6):e65378. doi: 10.1371/journal.pone.0065378. Print 2013. PMID 23762355
- [Background] Lee CS, Kang KC, Chung SS, Park WH, Shin WJ, Seo YG. How does back muscle strength change after posterior lumbar interbody fusion? J Neurosurg Spine. 2017 Feb;26(2):163-170. doi: 10.3171/2016.7.SPINE151132. Epub 2016 Oct 14. PMID 27740397
- [Background] Mancuso CA, Reid MC, Duculan R, Girardi FP. Improvement in Pain After Lumbar Spine Surgery: The Role of Preoperative Expectations of Pain Relief. Clin J Pain. 2017 Feb;33(2):93-98. doi: 10.1097/AJP.0000000000000383. PMID 27022672
- [Background] Mannion AF, Porchet F, Kleinstuck FS, Lattig F, Jeszenszky D, Bartanusz V, Dvorak J, Grob D. The quality of spine surgery from the patient's perspective. Part 1: the Core Outcome Measures Index in clinical practice. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):367-73. doi: 10.1007/s00586-009-0942-8. Epub 2009 Mar 25. PMID 19319578